CLINICAL TRIAL: NCT06424769
Title: Improving Outcomes and Reducing Disparities for Patients With Inflammatory Bowel Disease Through Epidemiology and Enhanced Disease Management (PROMOTE IBD)
Brief Title: Improving Outcomes and Reducing Disparities for Patients With Inflammatory Bowel Disease Through Epidemiology and Enhanced Disease Management
Acronym: PROMOTE IBD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Pennsylvania (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-0699; 855107 (Other: University of Pennsylvania)
Record Dates: First submitted 2024-05-13; First posted 2024-05-22 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Colitis
Keywords: Text Messaging; Symptom Monitoring; Social Risk Factors
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Colitis | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: After completing their baseline survey, consented participants will be randomized to usual care and intervention groups in a 2:1 allocation ratio. A computer-generated, centralized randomization with permuted block randomization within sites to ensure allocation concealment will be utilized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Digital Care Arm (Active Comparator): Participants will receive brief check-in surveys about their IBD symptoms minimally once a month, via text messaging. Participants will also receive IBD educational text messages twice each week.
  Interventions: Other: Enhanced Digital Care; Other: Education
- Specialized Education Arm (Placebo Comparator): Participants in this arm will receive IBD educational text messages twice each week.
  Interventions: Other: Education

INTERVENTIONS:
Other: Enhanced Digital Care — Participants will receive brief check-in surveys about their IBD symptoms once a month, via text messaging. If the survey response indicates significant symptoms, an alert will be sent to the participant's IBD care team and participant will receive more frequent surveys (weekly) over the next month. Participants and their IBD clinical team will be able to communicate by text for non-emergency IBD-related questions.
  Arms: Enhanced Digital Care Arm
Other: Education — Participants will receive education texts about IBD from trusted sources approximately twice a week. Topics will include: diet, medication adherence, fatigue, preventative care and other relevant issues.

SUMMARY:
The goal of this clinical trial is to learn whether IBD patients have better disease outcomes and feel more empowered to manage their condition if they have access to text messaging with their clinical team and if their symptoms are more regularly monitored through text-based surveys.

Researchers will compare participants who have access to text-based monitoring, communication and education to participants who have access to text-based education alone. Researchers will also examine if different social and other non-medical factors impact IBD symptoms and quality of life.

All participants will:

* complete 5 brief on-line surveys over 12 months about their IBD and social risk factors,
* receive IBD education content by text message up to 2 times a week.

Some participants will also:

* receive additional surveys by text to monitor their IBD progression,
* have the opportunity to directly text message their IBD medical team.

DETAILED DESCRIPTION:
Crohn's disease (CD) and ulcerative colitis (UC), collectively referred to as inflammatory bowel diseases (IBD), are chronic diseases with no cure. Patient activation, defined as having the knowledge, skill, and confidence to manage one's health, can improve outcomes in chronic diseases, including IBD. Tailored digital health interventions can facilitate proactive longitudinal care for IBD patients by improving patient activation, promoting self-management and remote monitoring and can be automated and implemented at scale.

The researchers are conducting a multi-center, open-label, randomized clinical trial to evaluate the effectiveness of a tailored digital health intervention versus usual care to improve disease management and patient activation among teenage and adult patients with IBD. The researchers hypothesize the intervention will lead to higher patient activation, improved outcomes and quality of life and reduced health disparities among children and adults with IBD. Within the usual care arm, researchers will measure Social Determinants of Health at enrollment and evaluate associations between these factors and time spent in remission over a 1-year follow-up period.

Participants in both arms will complete electronic surveys at baseline and then quarterly thereafter for 12-months. The baseline survey will include: 1) basic demographic information, 2) social risk assessment (adapted from the Health-related Social Needs Screening Tool by the Centers for Medicare & Medicaid Services (CMS) and the Centers for Disease Control and Prevention (CDC) National Health Interview Survey (NHIS) survey, this measure will be completed by the parent/guardian for pediatric participants), 3) patient reported outcomes for ulcerative colitis and Crohn's disease (PRO-2-UC or PRO-2-CD), 4) IBD-related quality of life (Short Inflammatory Bowel Disease Questionnaire (SIBDQ)), 5) IBD-related healthcare utilization, 6) IBD-related medication adherence and 7) patient activation measure (PAM Survey). All of these except demographic questions will be repeated at 12 months. Quarterly surveys at 3, 6, and 9 months will only include questions on IBD patient-reported outcomes and unplanned healthcare utilization (~8 questions) with the addition of medication adherence questions and the PAM at 6-months (12 additional questions).

In addition to these patient-reported data, providers and research coordinator at each site will perform chart abstraction to identify specific clinical disease-level factors (including disease severity and phenotype) and treatment-level factors (prior and current therapies).

Participants in both arms will receive texts approximately twice a week containing curated educational content. All participants will receive usual clinical care per discretion of their treating provider and will maintain usual healthcare interactions with the clinical team using their preferred method of interaction including phone or electronic communications within their Electronic Health Record (EHR).

Participants assigned to the intervention arm will receive enhanced electronic health care delivered through text messaging. This includes short monthly check in surveys to assess IBD disease progression. Survey cadence will increase to weekly for 4 weeks at a time if a participant reports severe symptoms. This also includes the opportunity to communicate with their clinical team through text messaging.

Among participants assigned to the usual care arm of the pragmatic trial, a cohort analysis will evaluate associations between social risk and IBD natural history and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 13+ years old with IBD (Crohn's disease, ulcerative colitis, indeterminant colitis).
* Followed at a participating site with an office visit (in-person or virtual) within the preceding 12 months.
* Have access to a mobile phone and willing and able to receive and respond to text messages.
* Willing to answer questions on electronic surveys.
* Have the ability to read text messages and answer surveys in English or Spanish.

Exclusion Criteria:

* IBD patients s/p surgery with a current pouch or ostomy.
* Unable to provide informed consent and child assent for minors.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Activation using PAM | Baseline, 12 months
  The primary outcome is the change in patient activation from baseline, with a 4-point improvement on Patient Activation Measure (PAM) scale considered a minimal clinically important difference (MCID). Patient activation is an assessment of the knowledge, skills and confidence of patients to manage their health. In chronic diseases, activated patients are more likely to adhere to treatment, perform regular self-monitoring at home and obtain regular chronic care. Activated patients are also more likely to make healthier lifestyle choices and preventative behaviors. Longitudinal improvement in patient activation measures is associated with improved clinical outcomes, decreased unplanned healthcare utilization and lower costs.

SECONDARY OUTCOMES:
Remission at 52 Weeks | 12 months
  Proportion of participants achieving Patient Reported Outcome (PRO) remission without steroids at end of study (among participants with active disease at baseline). This will be assessed for ulcerative colitis patients based on the 2-point PRO2-UC and assessed for Crohn's disease patients using the 2-point PRO2-CD. The PRO2-UC consists of the stool frequency and rectal bleeding subscores of the Mayo Clinic Score, and remission is defined as absence of rectal bleeding (rectal bleeding score = 0) and normal or near normal stool frequency (stool frequency score ≤1). The PRO2-CD consists of the 2 Crohn's Disease Activity Index (CDAI) component items: daily stool frequency and abdominal pain, and remission is defined as mean daily score of abdominal pain score ≤1 and stool frequency score ≤3.
IBD-Related Quality of Life | up to 12 months
  IBD-related quality of life will be measured using the Short Inflammatory Bowel Disease Questionnaire (SIBDQ), a validated, 10-item questionnaire which measures quality of life across physical, social and emotional domains in patients with IBD. The score on this questionnaire ranges from 10 to 70, with a minimal clinically important difference (MCID) of 9 points. This will be measured at baseline and at 12 months.
Unplanned Healthcare Utilization | up to 12 months
  Unplanned healthcare utilization (defined as IBD-related Emergency Department (ED) visit, hospitalization, or abdominal/perianal surgery for IBD) will be measured by self-report every 3 months (Baseline and months 3, 6, 9, and 12).

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Kappelman, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (8):
- United States (8):
  - University of California San Diego, San Diego, California
  - University of California San Francisco Benioff Children's Hospital, San Francisco, California
  - Morehouse School of Medicine, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - NYU Langone Health Lake Success, Lake Success, New York
  - UNC-Chapel Hill School of Medicine, Chapel Hill, North Carolina
  - Atrium Health Levine Children's, Charlotte, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: From 9 months after the end of the trial and publication of study results to up to 36 months.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Dahlhamer JM, Zammitti EP, Ward BW, Wheaton AG, Croft JB. Prevalence of Inflammatory Bowel Disease Among Adults Aged >/=18 Years - United States, 2015. MMWR Morb Mortal Wkly Rep. 2016 Oct 28;65(42):1166-1169. doi: 10.15585/mmwr.mm6542a3. PMID 27787492
- [Background] Singh S, Qian AS, Nguyen NH, Ho SKM, Luo J, Jairath V, Sandborn WJ, Ma C. Trends in U.S. Health Care Spending on Inflammatory Bowel Diseases, 1996-2016. Inflamm Bowel Dis. 2022 Mar 2;28(3):364-372. doi: 10.1093/ibd/izab074. PMID 33988697
- [Background] Baumgart DC, Le Berre C. Newer Biologic and Small-Molecule Therapies for Inflammatory Bowel Disease. N Engl J Med. 2021 Sep 30;385(14):1302-1315. doi: 10.1056/NEJMra1907607. No abstract available. PMID 34587387
- [Background] Liu JJ, Abraham BP, Adamson P, Barnes EL, Brister KA, Damas OM, Glover SC, Hooks K, Ingram A, Kaplan GG, Loftus EV, McGovern DPB, Narain-Blackwell M, Odufalu FD, Quezada S, Reeves V, Shen B, Stappenbeck TS, Ward L. The Current State of Care for Black and Hispanic Inflammatory Bowel Disease Patients. Inflamm Bowel Dis. 2023 Feb 1;29(2):297-307. doi: 10.1093/ibd/izac124. PMID 35816130
- [Background] Afzali A, Cross RK. Racial and Ethnic Minorities with Inflammatory Bowel Disease in the United States: A Systematic Review of Disease Characteristics and Differences. Inflamm Bowel Dis. 2016 Aug;22(8):2023-40. doi: 10.1097/MIB.0000000000000835. PMID 27379446
- [Background] Barnes EL, Loftus EV Jr, Kappelman MD. Effects of Race and Ethnicity on Diagnosis and Management of Inflammatory Bowel Diseases. Gastroenterology. 2021 Feb;160(3):677-689. doi: 10.1053/j.gastro.2020.08.064. Epub 2020 Oct 21. PMID 33098884
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Hibbard JH, Greene J. What the evidence shows about patient activation: better health outcomes and care experiences; fewer data on costs. Health Aff (Millwood). 2013 Feb;32(2):207-14. doi: 10.1377/hlthaff.2012.1061. PMID 23381511
- [Background] Anderson G, Rega ML, Casasanta D, Graffigna G, Damiani G, Barello S. The association between patient activation and healthcare resources utilization: a systematic review and meta-analysis. Public Health. 2022 Sep;210:134-141. doi: 10.1016/j.puhe.2022.06.021. Epub 2022 Aug 12. PMID 35970015
- [Background] Barnes EL, Long MD, Kappelman MD, Martin CF, Sandler RS. High Patient Activation Is Associated With Remission in Patients With Inflammatory Bowel Disease. Inflamm Bowel Dis. 2019 Jun 18;25(7):1248-1254. doi: 10.1093/ibd/izy378. PMID 30590700
- [Background] Haj O, Lipkin M, Kopylov U, Sigalit S, Magnezi R. Patient activation and its association with health indices among patients with inflammatory bowel disease. Therap Adv Gastroenterol. 2022 Oct 6;15:17562848221128757. doi: 10.1177/17562848221128757. eCollection 2022. PMID 36225610